CLINICAL TRIAL: NCT00003242
Title: An Open-Label, Non-Randomized Phase I Study of the Protein Kinase C Inhibitor Bryostatin-1 Administered in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Bryostatin 1 Plus Paclitaxel and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-139; CDR0000066117 (Registry Identifier: PDQ (Physician Data Query)); NCI-T97-0118
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — bryostatin 1; Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: bryostatin 1
Drug: cisplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy with bryostatin 1 plus paclitaxel and cisplatin in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of intravenous bryostatin 1 when administered in combination with a fixed dose of paclitaxel and cisplatin in patients with advanced solid tumors. II. Investigate the clinical pharmacokinetics of intravenous paclitaxel when administered in combination with bryostatin 1 in these patients. III. Obtain preliminary data on the therapeutic activity of this therapy in these patients and evaluate surrogate markers of activity.

OUTLINE: This is an open label, dose escalation study. Patients receive paclitaxel IV over 1 hour on day 1. On day 2, patients receive bryostatin 1 IV over 1 hour immediately followed by cisplatin IV on day 2. Treatment is repeated weekly for 3 consecutive weeks followed by one week of rest for at least 2 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are entered at escalating dose levels of bryostatin 1 and paclitaxel. If 2 of 6 patients experience dose limiting toxicity (DLT) at any given dose level, then the maximum tolerated dose (MTD) is declared to be the preceding dose level. Once the MTD of paclitaxel and bryostatin 1 has been established, escalations of weekly cisplatin will be added. Additional patient cohorts receive two escalating doses of paclitaxel and cisplatin with the fixed bryostatin 1 dose level, in the absence of DLT. Patients at a lower bryostatin 1 dose may be escalated to a higher bryostatin 1 dose, only if that higher dose has been proven to be safe in another cohort of patients.

PROJECTED ACCRUAL: An anticipated 3 to 60 patients will be accrued for this study within 1-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor Must be refractory to standard therapy or no standard therapy exists No CNS metastases or CNS primary malignancy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No history of cardiac arrhythmias No congestive heart failure No myocardial infarction in the last 6 months Neurologic: No grade 3 or greater neurotoxicity Other: HIV negative No serious or uncontrolled infection Not pregnant Adequate contraception required of all fertile patients during study and until 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: At least 6 weeks since prior nitrosoureas or mitomycin At least 4 weeks since other prior chemotherapy Must have recovered from prior chemotherapy Endocrine therapy: Must have recovered from prior endocrine therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-02; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States